CLINICAL TRIAL: NCT02140320
Title: A Randomised, Double Blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Treatment With Single and Repeat Doses of Inhaled RV1729 in Healthy Subjects for up to 28 Days and Subjects With Stable Asthma for 14 Days
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of RV1729 for up to 28 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STN003; 2014-000090-39 (EudraCT Number)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Asthma; Healthy Volunteers
MeSH Terms: conditions — Asthma | interventions — 6-(2-((4-amino-3-(3-hydroxyphenyl)-1H-pyrazolo(3,4-d)pyrimidin-1-yl)methyl)-3-(2-chlorobenzyl)-4-oxo-3,4-dihydroquinazolin-5-yl)-N,N-bis(2-methoxyethyl)hex-5-ynamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single dose (healthy volunteers) (Experimental)
  Interventions: Drug: RV1729 single dose; Drug: RV1729 matching placebo single dose
- 14 day repeat dose (healthy volunteers) (Experimental)
  Interventions: Drug: RV1729 14 day repeat dose; Drug: RV1729 matching placebo 14 day repeat dose
- 14 day repeat dose (asthma patients) (Experimental)
  Interventions: Drug: RV1729 14 day repeat dose; Drug: RV1729 matching placebo 14 day repeat dose
- 28 day repeat dose (healthy volunteers) (Experimental)
  Interventions: Drug: RV1729 28 day repeat dose; Drug: RV1729 matching placebo 28 day repeat dose

INTERVENTIONS:
Drug: RV1729 single dose — Safety and tolerability of single dose
  Arms: Single dose (healthy volunteers)
Drug: RV1729 matching placebo single dose — Safety and tolerability of single dose
  Arms: Single dose (healthy volunteers)
Drug: RV1729 14 day repeat dose — Safety and tolerability of repeat doses
  Arms: 14 day repeat dose (asthma patients); 14 day repeat dose (healthy volunteers)
Drug: RV1729 matching placebo 14 day repeat dose — Safety and tolerability of repeat doses
  Arms: 14 day repeat dose (asthma patients); 14 day repeat dose (healthy volunteers)
Drug: RV1729 28 day repeat dose — Safety and tolerability of repeat doses
  Arms: 28 day repeat dose (healthy volunteers)
Drug: RV1729 matching placebo 28 day repeat dose — Safety and tolerability of repeat doses
  Arms: 28 day repeat dose (healthy volunteers)

SUMMARY:
RV1729 is a new medicine being developed for the potential treatment of asthma and smoking related lung disease (also known as chronic obstructive pulmonary disease - COPD).

The objective of this study is to investigate the safety, tolerability and pharmacokinetics of single doses of RV1729 and repeat doses of RV1729 for up to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Be a man or woman between 18 to 60 years of age, inclusive, at the time of signing the informed consent.
* Cohorts 1, 2 & 3 women of childbearing potential must have a documented menstrual period prior to the first dose and be willing to use 2 forms of appropriate methods of contraception from screening until 4 months after the final dose of RV1729, OR
* Women of non-childbearing potential must be spontaneously amenorrhoeic for at least 1 year or have been permanently sterilised, OR
* If a man, must be willing and able to use one of the contraception methods listed in the protocol and agree not to donate sperm from screening until 4 months after the final dose of RV1729
* Women must agree not to donate eggs (ova, oocytes) from screening until at least 6 months after the final dose of RV1729
* Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Body mass index between 19 and 30 kg/m2 and body weight not less than 50 kg.
* Vital sign assessments within normal ranges
* Have a 12-lead ECG recording consistent with normal cardiac function
* Capable of complying with all study restrictions and procedures including ability to use the study inhaler correctly

Cohorts 1, 2 & 4 (healthy volunteers only)

* Healthy as determined by a physician, based on a full medical evaluation including medical history, physical examination and laboratory tests.
* Pre-bronchodilator spirometry readings (FEV1 and FVC) to be ≥80% predicted value and FEV1/FVC ratio >0.7
* Not taking prescription medications for 14 days prior to screening and agree not to use prescription medications throughout the duration of the study (with the exception of the use of contraceptives or hormone replacement therapy).
* Not taking over-the-counter medications and herbal medication for 14 days prior to screening throughout the study.

Cohort 3 (asthma patients only)

* Documented history of asthma, at least 6 months prior to screening and currently being treated with daily inhaled corticosteroids with or without long acting beta-agonist (LABA)
* Have a diagnosis of asthma. This will be confirmed by bronchodilator reversibility at screening
* Have a pre-bronchodilator FEV1 ≥60% and ≤85% of predicted normal value
* Have stable asthma based with no exacerbation requiring change in therapy for 12 weeks and no hospitalisation or visit to accident and emergency for asthma in the 12 months prior to screening.
* Not have a clinical abnormality or laboratory parameters outside the reference range.
* Not taking prescription medications for 14 days prior to screening and agree not to use prescription medications throughout the duration of the study except for use of contraceptives or hormone replacement therapy and treatment for asthma
* Not taking over-the-counter medications and herbal medication for 14 days, or antihistamines for 7 days prior to the screening visit and agree to refrain from taking such medications throughout the study.

Exclusion Criteria:

* Upper or lower respiratory tract infection within 4 weeks before screening
* Clinically significant abnormal values for haematology, clinical chemistry or urinalysis at screening or Day -1
* Has a history of or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease.
* History of, or a reason to believe a subject has a history of drug or alcohol abuse within the past 5 years.
* Positive test for alcohol or drugs of abuse, including cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines or barbiturates at screening or on Day -1
* History of clinically significant allergies that, in the opinion of the Investigator or Medical Monitor, would contraindicate their participation.
* Subjects known to suffer from hayfever, or other allergy, that may require antihistamine therapy during the course of the study.
* Known allergy to the study drug or any of the excipients of the formulation or has previously been exposed to RV1729.
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months or intention to donate blood or blood products during the study.
* Received an experimental drug or used an experimental medical device within 3 months or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled.
* If a woman has a positive serum pregnancy test at screening or a positive urine pregnancy test on Day -1, is pregnant, breast-feeding or planning to become pregnant during the study.
* Liver function test results >1.5 x ULN (upper limit of normal) at Screening or on Day -1.
* Positive test for human immunodeficiency virus (HIV) 1 and 2 antibodies, hepatitis B virus (HBV) infection or hepatitis C antibodies.
* History of smoking or use of nicotine-containing substances within the previous 6 months, or a positive carbon monoxide test at screening or on Day -1 (or a smoking history ≥ 10 pack years).
* Preplanned surgery or procedures that would interfere with the conduct of the study.
* Employee of the Investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that Investigator or study centre, as well as family members of the employees or the Investigator.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study.
* The subject is unable or unwilling to comply fully with the study protocol.
* Subject is mentally or legally incapacitated.
* Unable or unwilling to undergo multiple venepuncture procedures or the subject has poor access to veins suitable for cannulation.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Cohorts 1, 2 & 4 (healthy volunteers only)

* Any chronic illness or clinically relevant abnormality identified on the screening medical assessment, laboratory tests or ECG

Cohort 3 (asthma patients only)

* Administration of oral, injectable or dermal steroids or leukotriene modifiers within 3 months or intranasal steroids within 1 week of the screening visit.
* Has ever had an episode of life-threatening asthma defined as respiratory arrest, intubation for asthma, or intensive care unit admission for asthma.
* Any acute or chronic illness or clinically relevant abnormality other than asthma identified on the screening medical assessment, laboratory tests or ECG.
* Has severe asthma based on Investigator assessment and/or use of prohibited asthma medications.

Cohort 4 (healthy volunteers only)

* Women of child bearing potential

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Cohort 1, 56 days: Cohorts 2 & 3, 70 days: Cohort 4, 84 days
  Assessment of the number of adverse events reported by subjects following dosing
ECG assessment (12-lead ECG) | Cohort 1, 29 days: Cohorts 2 & 3, 42 days: Cohort 4, 56 days
  Change from pre-dose values
Vital sign assessment (blood pressure and heart rate, measured together) | Cohort 1, 29 days: Cohorts 2 & 3, 42 days: Cohort 4, 56 days
  Change from pre-dose values
Clinical laboratory assessments (blood and urine samples, collected together) | Cohort 1, 29 days: Cohorts 2 & 3, 42 days: Cohort 4, 56 days
  Change from pre-dose values
Spirometry assessment (FEV1 & FVC) | Cohort 1, 29 days: Cohorts 2 & 3, 42 days: Cohort 4, 56 days
  Change from pre-dose values

SECONDARY OUTCOMES:
Plasma RV1729 levels | Cohort 1: Day 1, 7 samples, Day 2-29, 5 samples; Cohorts 2 & 3: Days 1, 7 & 14, 8 samples, Days 2 & 8-13, 1 sample per day, Days 15-42, 6 samples; Cohort 4: Days 1, 14 & 28, 8 samples, Days 2, 7, 15, 21, 26 & 27, 1 sample per day, Days 29-70, 7 samples;

OTHER OUTCOMES:
Serum biomarkers (measuring markers of inflammation in the blood) | Cohort 2: Days 1 & 14, 2 samples per day, Days 2, 7, 15 & 42, 1 sample per day; Cohort 3: Days 1 & 14, 2 samples per day, Days 2, 7, 15, 21 & 42, 1 sample per day; Cohort 4: Days 1 & 14, 2 samples per day, Days 7, 21, 29 & 56, 1 sample per day;
Exhaled nitric oxide (measuring airway inflammation) | Cohort 3: Days 1 & 4 - 1 sample, Day 14 - 2 samples
Exhaled breath condensate (measuring markers of oxidate stress) | Cohort 3: Days 1 & 14 - 2 samples per day, Days 17 to 42 - 4 samples
Urinary cortisol and leukotriene E4 (LTE4) | Cohort 3: Days -1 & 14 (0 - 24 h collection)

CONTACTS AND LOCATIONS:
Overall Officials: Liza O'Dowd, MD, Study Director — Sponsor GmbH
Locations (2):
- United Kingdom (2):
  - London
  - Manchester